CLINICAL TRIAL: NCT06063109
Title: A Two-arm, Open-label, Single-sequence, Multiple Oral Dosings, Crossover Clinical Trial to Evaluate the Safety and the Pharmacokinetic Interaction of THP-00101 and THP-00102 in Healthy Adult Volunteers
Brief Title: A Clinical Trial to Evaluate the Safety and the Pharmacokinetic Interaction of Telmisartan and Dapagliflozin.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: THPharm Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THP-001-001
Record Dates: First submitted 2023-09-08; First posted 2023-10-02 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-09

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Telmisartan

STUDY DESIGN:
Intervention Model Description: A two-arm, open-label, single-sequence, multiple oral dosings, crossover clinical trials
  THP-00101 (Dapagliflozin) 10mg (18 Subjects): Tx A (5 days) -> Tx B (5 days) Treatment A: THP-00101 (Dapagliflozin) 10mg/5 days Treatment B: THP-00101 (Dapagliflozin) 10mg/5 days + THP-00102 (Telmisartan) 80mg/5 days
  THP-00102 (Telmisartan) 80mg (32 Subjects): Tx C (5 days) -> Tx B (5 days) Treatment C: THP-00102 (Telmisartan) 80mg/5 days Treatment B: THP-00102 (Telmisartan) 80mg/5 days + THP-00101 (Dapagliflozin) 10mg/5 days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): THP-00101 (Dapagliflozin) 10mg (18 Subjects): Tx A (5 days) -> Tx B (5 days) Treatment A: THP-00101 (Dapagliflozin) 10mg/5 days Treatment B: THP-00101 (Dapagliflozin) 10mg/5 days + THP-00102 (Telmisartan) 80mg/5 days
  Interventions: Drug: THP-00101 (Dapagliflozin) 10mg; Drug: THP-00102 (Telmisartan) 80mg
- Telmisartan (Experimental): THP-00102 (Telmisartan) 80mg (32 Subjects): Tx C (5 days) -> Tx B (5 days) Treatment C: THP-00102 (Telmisartan) 80mg/5 days Treatment B: THP-00102 (Telmisartan) 80mg/5 days + THP-00101 (Dapagliflozin) 10mg/5 days
  Interventions: Drug: THP-00101 (Dapagliflozin) 10mg; Drug: THP-00102 (Telmisartan) 80mg

INTERVENTIONS:
Drug: THP-00101 (Dapagliflozin) 10mg — Dapagliflozin 10mg Tablet / 5 days in period 1 and period 2 will be given to Arm A Dapagliflozin 10mg Tablet / 5 days in period 2 will be given to Arm B
  Other Names: Forxiga Tab. 10mg
Drug: THP-00102 (Telmisartan) 80mg — Telmisartan 80mg Tablet / 5 days in period 1 and period 2 will be given to Arm B Telmisartan 80mg Tablet / 5 days in period 2 will be given to Arm A
  Other Names: Micardis Tab. 80mg

SUMMARY:
The study was designed to evaluate the safety and pharmacokinetic interaction between THP-00101 and THP-00102 in healthy adult volunteers.

DETAILED DESCRIPTION:
The study consists of 2 periods of THP-00101 or THP00102 administration over 5 days and combined administration of THP-00101 and THP00102 over 5 days in two arms.

Dapagliflozin (18 Subjects): Tx A (5 days) -> Tx B (5 days) Treatment A: THP-00101 (Dapagliflozin) 1 tablet/5 days Treatment B: THP-00101 (Dapagliflozin) 1 tablet/5 days + THP-00102 (Telmisartan) 1 tablet/5 days

Telmisartan (32 Subjects): Tx C (5 days) -> Tx C (5 days) Treatment C: THP-00102 (Telmisartan) 1 tablet/5 days Treatment B: THP-00102 (Telmisartan) 1 tablet/5 days + THP-00101 (Dapagliflozin) 1 tablet/5 days

ELIGIBILITY:
Inclusion Criteria:

1. A person who is 19 years of age or older at the screening visit
2. A person who weighs at least 55 kg (50 kg for women) and has a body mass index (BMI) of at least 18.0 kg/m2 and at least 30.0 kg/m2 at screening visit

   ☞ BMI (kg/m2) = Weight (kg)/ {Height (m)}2
3. A person who has no clinically meaningful congenital or chronic disease and has no pathological symptoms or findings as a result of medical examination at a screening visit
4. A person who has been determined to be suitable for the test as a result of diagnostic tests such as hematology tests, hematochemical tests, serum tests, urine tests, etc., set and conducted by the test manager (or delegated test doctor) according to the characteristics of clinical drugs
5. A person who agrees to exclude the possibility of pregnancy using a medically recognized contraceptive method* (except hormones) and does not provide sperm or eggs from the date of first administration of the clinical trial drug to 14 days after the date of last clinical trial drug administration

   *medically-accepted Contraceptive methods: a combination of intrauterine devices, vasectomy, tubular ligation, and blocking contraception (male condoms, female condoms, cervical caps, contraceptive septum, sponge, etc.) or a combination of two or more blocking contraceptives
6. A person who has received and understood sufficient explanation of the purpose, contents, characteristics of clinical trial drugs, expected abnormal cases, etc., and signed the consent form according to his/her free will

Exclusion Criteria:

1. A person who has or has a history of clinically significant diseases corresponding to the digestive system, cardiovascular system, endocrine system, respiratory system, blood and tumor, infectious disease, kidney and urinary system, mental and nervous system, musculoskeletal system
2. A person who has a history of gastrointestinal surgery (excluding simple appendectomy or hernia surgery) or has gastrointestinal diseases that may affect drug absorption
3. Those who have taken drug metabolism-inducing and inhibiting drugs such as barbital drugs within one month of the first administration date, or drugs that may interfere with this clinical trial within 10 days of the first administration (however, in consideration of pharmacokinetic and pharmacokinetic characteristics of combination drugs it may consider as possible)
4. A person who participates in other clinical trials or biological equivalence tests within six months of the first administration and administered clinical trial drugs
5. A person who has donated whole blood within 8 weeks of the first administration, donated ingredients within 2 weeks or received a blood transfusion within 4 weeks from the first administration
6. A person who meets the following conditions within one month of the first dose date

   * Men consume an average of 21 cups/week of alcohol
   * Women consume an average of 14 cups/week of alcohol

     (1 glass = 50mL of soju, 30mL of spirits, or 250mL of beer)
   * An average of more than 20 cigarettes a day
7. A patient who falls under the following

   * Patients with a history of hypersensitivity to the main ingredient or additive of this drug
   * Type 1 diabetes patient with diabetic ketoacidosis
   * Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
   * A patient on dialysis
   * Patients with severe liver disorders, biliary obstruction, or bile congestion (mostly this drug is excreted as bile). A decrease in liver cleaning rate can be expected in patients with bile congestion, biliary obstruction disease, or liver failure.)
   * Patients with hereditary angioedema, or patients with a history of angioedema when treated with ACE inhibitors or angiotensin II receptor antagonists
   * Combination with aliskiren-containing preparations in patients with diabetes or moderate to severe renal disabilities (glomerular filtration rate <60mL/min/1.73m2)
8. For reasons other than the above selection and exclusion criteria, the person in charge of testing (or the delegated test doctor) determines that he/she is not suitable for participation in this clinical trial
9. In the case of female volunteers, those suspected of being pregnant or nursing

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - AUCτ,ss | Day 1 to Day 11
  AUCτ,ss of Dapagliflozin & Telmisartan
Pharmacokinetics - Cmax,ss | Day 1 to Day 11
  Cmax,ss of Dapagliflozin & Telmisartan
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Day 1 to Day 17
  Evaluate incidents rate of Adverse Event of Treatment-Emergent Adverse Event and compare concomitant medication usage

SECONDARY OUTCOMES:
Pharmacokinetics - Tmax,ss | Day 1 to Day 11
  Tmax,ss of Dapagliflozin & Telmisartan
Pharmacokinetics - Cmin,ss | Day 1 to Day 11
  Cmin,ss of Dapagliflozin & Telmisartan
Pharmacokinetics - CLss/F | Day 1 to Day 11
  CLss/F of Dapagliflozin & Telmisartan
Pharmacokinetics - Vdss/F | Day 1 to Day 11
  Vdss/F of Dapagliflozin & Telmisartan
Pharmacokinetics - PTF | Day 1 to Day 11
  Peak-trough Fluctuation of Dapagliflozin & Telmisartan

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hyun Kang, M.D, Principal Investigator — H Plus Yangji Hospital
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No